CLINICAL TRIAL: NCT03353597
Title: Reversing Epigenetic & Other Markers of Senescence by Transfusing Young Plasma To Older Human Subjects
Acronym: RESET-YOUTH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chandra Duggirala (Industry)
Responsible Party: Sponsor-Investigator, Chandra Duggirala, Principal Investigator, Fountain Labs, Inc.
Organization: Fountain Labs, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFP-1
Record Dates: First submitted 2017-11-07; First posted 2017-11-27 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Plasma Transfusion (Experimental): Plasma Transfusions with 2 units of plasma per dose, for a total of 6 doses
  Interventions: Biological: Plasma Transfusion

INTERVENTIONS:
Biological: Plasma Transfusion — All subjects will receive monthly, 2-unit transfusions of young healthy male donor plasma for total of 6 treatments. The plasma will be administered at a transfusion services facility in a manner consistent with generally accepted and standard guidelines for plasma transfusions.

SUMMARY:
This trial is designed to study the effects of monthly transfusions of young healthy male donor plasma on biological age as assessed by DNA methylation levels, and changes in cognitive, renal, and pulmonary function, muscle strength, telomere length, testosterone, estrogen, DHEAS, IGF-1, high resolution C-Reactive protein, and expression of P16INK4a in peripheral blood T lymphocytes and skin biopsies.

DETAILED DESCRIPTION:
Aging is a process for which there is no cure. Plasma transfusions, based on extensive animal studies, have the potential to reverse many, systemic age-related changes in the human body as well as age related chronic diseases. This is a non-randomized, uncontrolled phase I/II study to study the effects of monthly transfusions of young healthy male donor plasma on biological age as assessed by DNA methylation levels, and changes in cognitive, renal, and pulmonary function, muscle strength, telomere length, testosterone, estrogen, DHEAS, IGF-1, high resolution C-Reactive protein, and expression of p16INK4a in peripheral blood T lymphocytes and skin biopsies. To determine the safety and tolerability of monthly, 2-unit transfusions of young (<25 years of age) healthy male donor plasma for 6 months in patients older then 40 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40.
* Stable medications for 2 months prior to Screening.
* Signed and dated written informed consent obtained from the subject in accordance with local Institutional Review Board regulations.
* Males and all Women of Child Bearing Potential agree to abstain from sex or use an adequate method of contraception for the duration of the study and for 30 days after the last dose of study drug. Adequate contraceptive methods include those with a low failure rate, i.e., less than 1% per year, when used consistently and correctly), and , a woman who has been surgically sterilized or who has been in a state of amenorrhea.

Exclusion Criteria:

* Dementia of any etiology.
* Any medical condition other than dementia that could account for cognitive deficits (e.g., active seizure disorder, stroke, Central Nervous System diseases);
* History of significant cardiovascular, hematologic, renal, or advanced hepatic disease (or laboratory evidence thereof);
* History of major psychiatric illness or untreated depression;
* Neutrophil count <1,500/mm3, platelets <100,000/mm3, serum creatinine >1.5x upper limit of normal (ULN), total bilirubin >1.5 x ULN, Alanine Transaminase >3 x ULN, Aspartate Transaminase >3 x ULN, or International Normalized Ratio (INR) >1.2 at Screening evaluations;
* Evidence of any clinically significant findings on Screening or baseline evaluations which, in the opinion of the Investigator would pose a safety risk or interfere with appropriate interpretation of study data;
* Current or recent history (within four weeks prior to Screening) of a clinically significant bacterial, fungal, or mycobacterial infection;
* Current clinically significant viral infection;
* Major surgery within four weeks prior to Screening;
* Any contraindication to monthly plasma transfusions, including but not limited to:
* History of significant transfusion complications;
* Compatible plasma units not available;
* Prior intolerance to intravenous (IV) fluids;
* Immunoglobulin A deficiency by history or laboratory evidence at Screening;
* Bleeding;
* Any concurrent use of an anti-coagulant therapy.
* Daily administration of Aspirin 81mg will be allowed as long as the dose is stable for 30 days prior to Screening. Anti-platelet drugs are acceptable.
* Treatment with another investigational drug or participation in another interventional clinical trial within 3 months of Screening;
* Treatment with any human blood product, including IV immunoglobulin, during the 6 months prior to Screening or during the trial;
* Pregnant or lactating;
* Positive pregnancy test at Screening or Baseline (Day 1);
* Cancer within 5 years of Screening, except for nonmetastatic skin cancer or non-metastatic prostate cancer not expected to cause significant morbidity or mortality within one year of Baseline.
* AB blood type.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2120 (Estimated)
Dates: Start 2018-05-15 (Estimated); Primary Completion 2020-06-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Biological age as assessed by DNA methylation levels, to calculate the Epigenetic age. | Baseline to end of Month 9.
  The "epigenetic clock," as assessed by DNA methylation levels, which has been shown to be highly correlated with biologic age, longevity and is an independent predictor of mortality.

SECONDARY OUTCOMES:
Mental (Cognitive) Function | Baseline and Month 9
  Executive functioning, as measured by the California Stroop test
Lung (Pulmonary) Function | Baseline and Month 9
  FEV1 (Forced Expiratory Volume during the first second), and Peak Expiratory Flow
Kidney (Renal) Function | Baseline and Month 9
  Twenty-four hour urine collections will be performed by patients at Baseline and at Month 9. Creatinine Clearance, a measure of Renal function will be determined by calculating the glomerular filtration rate (GFR), which is the sum of filtration rates in all functioning nephrons.
Muscle Strength | Baseline and Month 9
  Unilateral Maximal Voluntary Isometric and Concentric Strength
Telomere Length | Baseline and Month 9
  A telomere is a region of repetitive nucleotide sequences at each end of a chromosome, which protects the end of the chromosome from deterioration or from fusion with neighboring chromosomes.
  Telomere shortening is associated with aging, mortality and aging-related diseases. Average telomere length will be measured in white blood cells by real time PCR technique.
Testosterone | Baseline and Month 9
  Serum free and total Testosterone levels
Estrogen | Baseline and Month 9
  Serum Estrogen levels
DHEAS | Baseline and Month 9
  Dehydroepiandrosterone is an endogenous steroid hormone that has a role in the synthesis of sex steroids (androgens and estrogens), as well as neurotrophic and other effects
IGF-1 | Baseline and Month 9
  Insulin Like Growth Factor -1(IGF-1) declines continuously with aging in adults, and has been shown to mediate a number of pathways that are associated with longevity.
High Sensitivity C-Reactive Protein | Baseline and Month 9
  C-Reactive Protein is a blood protein that is a marker of inflammation. Studies have suggested that a persistent level of inflammation plays a major role in cardiovascular and other degenerative and aging related diseases.
P16INK4a (A marker of cellular aging) | Baseline and Month 9
  The cyclin- dependent kinase inhibitor CDKN2A, commonly referred to as p16INK4a or p16, has been established as a general marker of cellular senescence or aging. The expression of p16INK4a has been shown to increase exponentially with chronologic age. P16-INK4a is performed on a small specimen of blood drawn from the subjects, as well as from skin biopsy samples.

OTHER OUTCOMES:
Exploratory biomarkers | Baseline,1,2,3,4,5,6, and 9 months.
  Blood, and urine, proteomic signatures of aging, including Interleukin-6, Tumor Necrosis Factor Alpha, Tissue Inhibitor of Metallo Proteinases-2, Transforming Growth Factor-Beta, and Mechanistic Target of Rapamycin (mTOR) levels, that are associated with various cellular, genetic and physiological mechanisms of aging will be measured at Baseline, 1,2,3,4,5,6, and 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chandra s duggirala, Principal Investigator — Fountain Labs, Inc.
Locations (1):
- The Infusion Center & Clinic, San Mateo, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alcedo J, Kenyon C. Regulation of C. elegans longevity by specific gustatory and olfactory neurons. Neuron. 2004 Jan 8;41(1):45-55. doi: 10.1016/s0896-6273(03)00816-x. PMID 14715134
- [Background] Apfeld J, Kenyon C. Regulation of lifespan by sensory perception in Caenorhabditis elegans. Nature. 1999 Dec 16;402(6763):804-9. doi: 10.1038/45544. PMID 10617200
- [Background] Baht GS, Silkstone D, Vi L, Nadesan P, Amani Y, Whetstone H, Wei Q, Alman BA. Exposure to a youthful circulaton rejuvenates bone repair through modulation of beta-catenin. Nat Commun. 2015 May 19;6:7131. doi: 10.1038/ncomms8131. PMID 25988592
- [Background] Baker DJ, Wijshake T, Tchkonia T, LeBrasseur NK, Childs BG, van de Sluis B, Kirkland JL, van Deursen JM. Clearance of p16Ink4a-positive senescent cells delays ageing-associated disorders. Nature. 2011 Nov 2;479(7372):232-6. doi: 10.1038/nature10600. PMID 22048312
- [Background] Baylin SB, Jones PA. A decade of exploring the cancer epigenome - biological and translational implications. Nat Rev Cancer. 2011 Sep 23;11(10):726-34. doi: 10.1038/nrc3130. PMID 21941284
- [Background] Bell JT, Tsai PC, Yang TP, Pidsley R, Nisbet J, Glass D, Mangino M, Zhai G, Zhang F, Valdes A, Shin SY, Dempster EL, Murray RM, Grundberg E, Hedman AK, Nica A, Small KS; MuTHER Consortium; Dermitzakis ET, McCarthy MI, Mill J, Spector TD, Deloukas P. Epigenome-wide scans identify differentially methylated regions for age and age-related phenotypes in a healthy ageing population. PLoS Genet. 2012;8(4):e1002629. doi: 10.1371/journal.pgen.1002629. Epub 2012 Apr 19. PMID 22532803
- [Background] Benayoun BA, Pollina EA, Brunet A. Epigenetic regulation of ageing: linking environmental inputs to genomic stability. Nat Rev Mol Cell Biol. 2015 Oct;16(10):593-610. doi: 10.1038/nrm4048. Epub 2015 Sep 16. PMID 26373265
- [Background] Bergman RJ, Gazit D, Kahn AJ, Gruber H, McDougall S, Hahn TJ. Age-related changes in osteogenic stem cells in mice. J Bone Miner Res. 1996 May;11(5):568-77. doi: 10.1002/jbmr.5650110504. PMID 9157771
- [Background] BLUEPRINT consortium. Quantitative comparison of DNA methylation assays for biomarker development and clinical applications. Nat Biotechnol. 2016 Jul;34(7):726-37. doi: 10.1038/nbt.3605. Epub 2016 Jun 27. PMID 27347756
- [Background] Bocklandt S, Lin W, Sehl ME, Sanchez FJ, Sinsheimer JS, Horvath S, Vilain E. Epigenetic predictor of age. PLoS One. 2011;6(6):e14821. doi: 10.1371/journal.pone.0014821. Epub 2011 Jun 22. PMID 21731603
- [Background] Bollati V, Schwartz J, Wright R, Litonjua A, Tarantini L, Suh H, Sparrow D, Vokonas P, Baccarelli A. Decline in genomic DNA methylation through aging in a cohort of elderly subjects. Mech Ageing Dev. 2009 Apr;130(4):234-9. doi: 10.1016/j.mad.2008.12.003. Epub 2008 Dec 27. PMID 19150625
- [Background] Brack AS, Conboy MJ, Roy S, Lee M, Kuo CJ, Keller C, Rando TA. Increased Wnt signaling during aging alters muscle stem cell fate and increases fibrosis. Science. 2007 Aug 10;317(5839):807-10. doi: 10.1126/science.1144090. PMID 17690295
- [Background] Brandli O, Schindler C, Kunzli N, Keller R, Perruchoud AP. Lung function in healthy never smoking adults: reference values and lower limits of normal of a Swiss population. Thorax. 1996 Mar;51(3):277-83. doi: 10.1136/thx.51.3.277. PMID 8779131
- [Background] Burch JB, Augustine AD, Frieden LA, Hadley E, Howcroft TK, Johnson R, Khalsa PS, Kohanski RA, Li XL, Macchiarini F, Niederehe G, Oh YS, Pawlyk AC, Rodriguez H, Rowland JH, Shen GL, Sierra F, Wise BC. Advances in geroscience: impact on healthspan and chronic disease. J Gerontol A Biol Sci Med Sci. 2014 Jun;69 Suppl 1(Suppl 1):S1-3. doi: 10.1093/gerona/glu041. PMID 24833579
- [Background] Burrows B, Lebowitz MD, Camilli AE, Knudson RJ. Longitudinal changes in forced expiratory volume in one second in adults. Methodologic considerations and findings in healthy nonsmokers. Am Rev Respir Dis. 1986 Jun;133(6):974-80. doi: 10.1164/arrd.1986.133.6.974. PMID 3717769
- [Background] Arai T, Yusa S, Kirimura K, Usami S. Cloning and sequencing of the cDNA encoding lipase I from Trichosporon fermentans WU-C12. FEMS Microbiol Lett. 1997 Jul 1;152(1):183-8. doi: 10.1111/j.1574-6968.1997.tb10426.x. PMID 9228786
- [Background] Campisi J, d'Adda di Fagagna F. Cellular senescence: when bad things happen to good cells. Nat Rev Mol Cell Biol. 2007 Sep;8(9):729-40. doi: 10.1038/nrm2233. PMID 17667954
- [Background] Castellano JM, Mosher KI, Abbey RJ, McBride AA, James ML, Berdnik D, Shen JC, Zou B, Xie XS, Tingle M, Hinkson IV, Angst MS, Wyss-Coray T. Human umbilical cord plasma proteins revitalize hippocampal function in aged mice. Nature. 2017 Apr 27;544(7651):488-492. doi: 10.1038/nature22067. Epub 2017 Apr 19. PMID 28424512
- [Background] Cawthon RM, Smith KR, O'Brien E, Sivatchenko A, Kerber RA. Association between telomere length in blood and mortality in people aged 60 years or older. Lancet. 2003 Feb 1;361(9355):393-5. doi: 10.1016/S0140-6736(03)12384-7. PMID 12573379
- [Background] Cawthon RM. Telomere length measurement by a novel monochrome multiplex quantitative PCR method. Nucleic Acids Res. 2009 Feb;37(3):e21. doi: 10.1093/nar/gkn1027. Epub 2009 Jan 7. PMID 19129229
- [Background] Chen BH, Marioni RE, Colicino E, Peters MJ, Ward-Caviness CK, Tsai PC, Roetker NS, Just AC, Demerath EW, Guan W, Bressler J, Fornage M, Studenski S, Vandiver AR, Moore AZ, Tanaka T, Kiel DP, Liang L, Vokonas P, Schwartz J, Lunetta KL, Murabito JM, Bandinelli S, Hernandez DG, Melzer D, Nalls M, Pilling LC, Price TR, Singleton AB, Gieger C, Holle R, Kretschmer A, Kronenberg F, Kunze S, Linseisen J, Meisinger C, Rathmann W, Waldenberger M, Visscher PM, Shah S, Wray NR, McRae AF, Franco OH, Hofman A, Uitterlinden AG, Absher D, Assimes T, Levine ME, Lu AT, Tsao PS, Hou L, Manson JE, Carty CL, LaCroix AZ, Reiner AP, Spector TD, Feinberg AP, Levy D, Baccarelli A, van Meurs J, Bell JT, Peters A, Deary IJ, Pankow JS, Ferrucci L, Horvath S. DNA methylation-based measures of biological age: meta-analysis predicting time to death. Aging (Albany NY). 2016 Sep 28;8(9):1844-1865. doi: 10.18632/aging.101020. PMID 27690265
- [Background] Christensen BC, Houseman EA, Marsit CJ, Zheng S, Wrensch MR, Wiemels JL, Nelson HH, Karagas MR, Padbury JF, Bueno R, Sugarbaker DJ, Yeh RF, Wiencke JK, Kelsey KT. Aging and environmental exposures alter tissue-specific DNA methylation dependent upon CpG island context. PLoS Genet. 2009 Aug;5(8):e1000602. doi: 10.1371/journal.pgen.1000602. Epub 2009 Aug 14. PMID 19680444
- [Background] Cohn NB, Dustman RE, Bradford DC. Age-related decrements in Stroop Color Test performance. J Clin Psychol. 1984 Sep;40(5):1244-50. doi: 10.1002/1097-4679(198409)40:53.0.co;2-d. PMID 6490922
- [Background] Conboy IM, Rando TA. Aging, stem cells and tissue regeneration: lessons from muscle. Cell Cycle. 2005 Mar;4(3):407-10. doi: 10.4161/cc.4.3.1518. Epub 2005 Mar 7. PMID 15725724
- [Background] Conboy IM, Conboy MJ, Wagers AJ, Girma ER, Weissman IL, Rando TA. Rejuvenation of aged progenitor cells by exposure to a young systemic environment. Nature. 2005 Feb 17;433(7027):760-4. doi: 10.1038/nature03260. PMID 15716955
- [Background] Conboy MJ, Conboy IM, Rando TA. Heterochronic parabiosis: historical perspective and methodological considerations for studies of aging and longevity. Aging Cell. 2013 Jun;12(3):525-30. doi: 10.1111/acel.12065. Epub 2013 Apr 10. PMID 23489470
- [Background] Conboy IM, Rando TA. The regulation of Notch signaling controls satellite cell activation and cell fate determination in postnatal myogenesis. Dev Cell. 2002 Sep;3(3):397-409. doi: 10.1016/s1534-5807(02)00254-x. PMID 12361602
- [Background] Conboy IM, Conboy MJ, Smythe GM, Rando TA. Notch-mediated restoration of regenerative potential to aged muscle. Science. 2003 Nov 28;302(5650):1575-7. doi: 10.1126/science.1087573. PMID 14645852
- [Background] Hernandez DG, Nalls MA, Gibbs JR, Arepalli S, van der Brug M, Chong S, Moore M, Longo DL, Cookson MR, Traynor BJ, Singleton AB. Distinct DNA methylation changes highly correlated with chronological age in the human brain. Hum Mol Genet. 2011 Mar 15;20(6):1164-72. doi: 10.1093/hmg/ddq561. Epub 2011 Jan 7. PMID 21216877
- [Background] Eggel A, Wyss-Coray T. A revival of parabiosis in biomedical research. Swiss Med Wkly. 2014 Feb 4;144:w13914. doi: 10.4414/smw.2014.13914. PMID 24496774
- [Background] Fraga MF, Esteller M. Epigenetics and aging: the targets and the marks. Trends Genet. 2007 Aug;23(8):413-8. doi: 10.1016/j.tig.2007.05.008. Epub 2007 Jun 7. PMID 17559965
- [Background] Gavrilov LA, Gavrilova NS. The reliability theory of aging and longevity. J Theor Biol. 2001 Dec 21;213(4):527-45. doi: 10.1006/jtbi.2001.2430. PMID 11742523
- [Background] Hannum G, Guinney J, Zhao L, Zhang L, Hughes G, Sadda S, Klotzle B, Bibikova M, Fan JB, Gao Y, Deconde R, Chen M, Rajapakse I, Friend S, Ideker T, Zhang K. Genome-wide methylation profiles reveal quantitative views of human aging rates. Mol Cell. 2013 Jan 24;49(2):359-367. doi: 10.1016/j.molcel.2012.10.016. Epub 2012 Nov 21. PMID 23177740
- [Background] Hortobagyi T, Zheng D, Weidner M, Lambert NJ, Westbrook S, Houmard JA. The influence of aging on muscle strength and muscle fiber characteristics with special reference to eccentric strength. J Gerontol A Biol Sci Med Sci. 1995 Nov;50(6):B399-406. doi: 10.1093/gerona/50a.6.b399. PMID 7583797
- [Background] Horvath S, Zhang Y, Langfelder P, Kahn RS, Boks MP, van Eijk K, van den Berg LH, Ophoff RA. Aging effects on DNA methylation modules in human brain and blood tissue. Genome Biol. 2012 Oct 3;13(10):R97. doi: 10.1186/gb-2012-13-10-r97. PMID 23034122
- [Background] Horvath S. DNA methylation age of human tissues and cell types. Genome Biol. 2013;14(10):R115. doi: 10.1186/gb-2013-14-10-r115. PMID 24138928
- [Background] Katsimpardi L, Litterman NK, Schein PA, Miller CM, Loffredo FS, Wojtkiewicz GR, Chen JW, Lee RT, Wagers AJ, Rubin LL. Vascular and neurogenic rejuvenation of the aging mouse brain by young systemic factors. Science. 2014 May 9;344(6184):630-4. doi: 10.1126/science.1251141. Epub 2014 May 5. PMID 24797482
- [Background] Jeong DE, Artan M, Seo K, Lee SJ. Regulation of lifespan by chemosensory and thermosensory systems: findings in invertebrates and their implications in mammalian aging. Front Genet. 2012 Oct 18;3:218. doi: 10.3389/fgene.2012.00218. eCollection 2012. PMID 23087711
- [Background] Kenyon C, Chang J, Gensch E, Rudner A, Tabtiang R. A C. elegans mutant that lives twice as long as wild type. Nature. 1993 Dec 2;366(6454):461-4. doi: 10.1038/366461a0. PMID 8247153
- [Background] Koch CM, Wagner W. Epigenetic-aging-signature to determine age in different tissues. Aging (Albany NY). 2011 Oct;3(10):1018-27. doi: 10.18632/aging.100395. PMID 22067257
- [Background] Krishnamurthy J, Torrice C, Ramsey MR, Kovalev GI, Al-Regaiey K, Su L, Sharpless NE. Ink4a/Arf expression is a biomarker of aging. J Clin Invest. 2004 Nov;114(9):1299-307. doi: 10.1172/JCI22475. PMID 15520862
- [Background] Li Y, Zhu J, Tian G, Li N, Li Q, Ye M, Zheng H, Yu J, Wu H, Sun J, Zhang H, Chen Q, Luo R, Chen M, He Y, Jin X, Zhang Q, Yu C, Zhou G, Sun J, Huang Y, Zheng H, Cao H, Zhou X, Guo S, Hu X, Li X, Kristiansen K, Bolund L, Xu J, Wang W, Yang H, Wang J, Li R, Beck S, Wang J, Zhang X. The DNA methylome of human peripheral blood mononuclear cells. PLoS Biol. 2010 Nov 9;8(11):e1000533. doi: 10.1371/journal.pbio.1000533. PMID 21085693
- [Background] Perna L, Zhang Y, Mons U, Holleczek B, Saum KU, Brenner H. Epigenetic age acceleration predicts cancer, cardiovascular, and all-cause mortality in a German case cohort. Clin Epigenetics. 2016 Jun 3;8:64. doi: 10.1186/s13148-016-0228-z. eCollection 2016. PMID 27274774
- [Background] Lei MK, Beach SR, Dogan MV, Philibert RA. A pilot investigation of the impact of smoking cessation on biological age. Am J Addict. 2017 Mar;26(2):129-135. doi: 10.1111/ajad.12502. Epub 2017 Jan 20. PMID 28106943
- [Background] Christiansen L, Lenart A, Tan Q, Vaupel JW, Aviv A, McGue M, Christensen K. DNA methylation age is associated with mortality in a longitudinal Danish twin study. Aging Cell. 2016 Feb;15(1):149-54. doi: 10.1111/acel.12421. Epub 2015 Nov 17. PMID 26594032
- [Background] Levine ME, Lu AT, Bennett DA, Horvath S. Epigenetic age of the pre-frontal cortex is associated with neuritic plaques, amyloid load, and Alzheimer's disease related cognitive functioning. Aging (Albany NY). 2015 Dec;7(12):1198-211. doi: 10.18632/aging.100864. PMID 26684672
- [Background] Liu Y, Sanoff HK, Cho H, Burd CE, Torrice C, Ibrahim JG, Thomas NE, Sharpless NE. Expression of p16(INK4a) in peripheral blood T-cells is a biomarker of human aging. Aging Cell. 2009 Aug;8(4):439-48. doi: 10.1111/j.1474-9726.2009.00489.x. Epub 2009 May 22. PMID 19485966
- [Background] Gorodinskii SM, Es'kova-Soskovets LS, Rokhlin MI, Sokolov IuIa, Turkin AD, Fishevskaia EA, Cherednichenko VA, Shatskii SN, Shorokhov AI. [A study of the absorption of vapors of I-131 compounds by the human skin]. Med Radiol (Mosk). 1967 Aug;12(8):57-60. No abstract available. Russian. PMID 5617346
- [Background] Marioni RE, Shah S, McRae AF, Chen BH, Colicino E, Harris SE, Gibson J, Henders AK, Redmond P, Cox SR, Pattie A, Corley J, Murphy L, Martin NG, Montgomery GW, Feinberg AP, Fallin MD, Multhaup ML, Jaffe AE, Joehanes R, Schwartz J, Just AC, Lunetta KL, Murabito JM, Starr JM, Horvath S, Baccarelli AA, Levy D, Visscher PM, Wray NR, Deary IJ. DNA methylation age of blood predicts all-cause mortality in later life. Genome Biol. 2015 Jan 30;16(1):25. doi: 10.1186/s13059-015-0584-6. PMID 25633388
- [Background] Kenyon CJ. The genetics of ageing. Nature. 2010 Mar 25;464(7288):504-12. doi: 10.1038/nature08980. PMID 20336132
- [Background] Rando TA. Stem cells, ageing and the quest for immortality. Nature. 2006 Jun 29;441(7097):1080-6. doi: 10.1038/nature04958. PMID 16810243
- [Background] Ruckh JM, Zhao JW, Shadrach JL, van Wijngaarden P, Rao TN, Wagers AJ, Franklin RJ. Rejuvenation of regeneration in the aging central nervous system. Cell Stem Cell. 2012 Jan 6;10(1):96-103. doi: 10.1016/j.stem.2011.11.019. PMID 22226359
- [Background] Stolzel F, Brosch M, Horvath S, Kramer M, Thiede C, von Bonin M, Ammerpohl O, Middeke M, Schetelig J, Ehninger G, Hampe J, Bornhauser M. Dynamics of epigenetic age following hematopoietic stem cell transplantation. Haematologica. 2017 Aug;102(8):e321-e323. doi: 10.3324/haematol.2016.160481. Epub 2017 May 26. No abstract available. PMID 28550187
- [Background] Wecker NS, Kramer JH, Wisniewski A, Delis DC, Kaplan E. Age effects on executive ability. Neuropsychology. 2000 Jul;14(3):409-14. doi: 10.1037//0894-4105.14.3.409. PMID 10928744
- [Background] Villeda SA, Plambeck KE, Middeldorp J, Castellano JM, Mosher KI, Luo J, Smith LK, Bieri G, Lin K, Berdnik D, Wabl R, Udeochu J, Wheatley EG, Zou B, Simmons DA, Xie XS, Longo FM, Wyss-Coray T. Young blood reverses age-related impairments in cognitive function and synaptic plasticity in mice. Nat Med. 2014 Jun;20(6):659-63. doi: 10.1038/nm.3569. Epub 2014 May 4. PMID 24793238
- [Background] Villeda SA, Luo J, Mosher KI, Zou B, Britschgi M, Bieri G, Stan TM, Fainberg N, Ding Z, Eggel A, Lucin KM, Czirr E, Park JS, Couillard-Despres S, Aigner L, Li G, Peskind ER, Kaye JA, Quinn JF, Galasko DR, Xie XS, Rando TA, Wyss-Coray T. The ageing systemic milieu negatively regulates neurogenesis and cognitive function. Nature. 2011 Aug 31;477(7362):90-4. doi: 10.1038/nature10357. PMID 21886162
- [Background] Thompson RF, Atzmon G, Gheorghe C, Liang HQ, Lowes C, Greally JM, Barzilai N. Tissue-specific dysregulation of DNA methylation in aging. Aging Cell. 2010 Aug;9(4):506-18. doi: 10.1111/j.1474-9726.2010.00577.x. Epub 2010 May 22. PMID 20497131
- [Background] Teschendorff AE, Menon U, Gentry-Maharaj A, Ramus SJ, Weisenberger DJ, Shen H, Campan M, Noushmehr H, Bell CG, Maxwell AP, Savage DA, Mueller-Holzner E, Marth C, Kocjan G, Gayther SA, Jones A, Beck S, Wagner W, Laird PW, Jacobs IJ, Widschwendter M. Age-dependent DNA methylation of genes that are suppressed in stem cells is a hallmark of cancer. Genome Res. 2010 Apr;20(4):440-6. doi: 10.1101/gr.103606.109. Epub 2010 Mar 10. PMID 20219944